CLINICAL TRIAL: NCT01647451
Title: A Randomised, Double-blind, Placebo-controlled, Parallel-group Trial to Assess Clinical Efficacy of NNC0114-0006 in Subjects With Active Rheumatoid Arthritis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NN8828-3842; 2011-005376-42 (EudraCT Number); U1111-1125-6552 (Other: WHO)
Record Dates: First submitted 2012-07-19; First posted 2012-07-23 (Estimated); Last update posted 2017-02-07 (Estimated); Status verified 2017-02

CONDITIONS: Inflammation; Rheumatoid Arthritis
MeSH Terms: conditions — Inflammation; Arthritis, Rheumatoid

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Active (Experimental)
  Interventions: Drug: NNC0114-0006
- Placebo (Placebo Comparator)
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: NNC0114-0006 — Two i.v. (intravenous) doses administered 6 weeks apart.
  Arms: Active
Drug: placebo — Two i.v. (intravenous) doses administered 6 weeks apart.
  Arms: Placebo

SUMMARY:
This trial is conducted in Europe. The aim of the trial is to evaluate the change in disease activity following intravenous (i.v.) administration of two doses of NNC0114-0006 compared to placebo in subjects with active rheumatoid arthritis (RA) on background methotrexate (MTX) therapy.

ELIGIBILITY:
Inclusion Criteria:

* A diagnosis of RA meeting the 2010 ACR (American College of Rheumatology) classification criteria, obtained at least 6 months prior to dosing with the trial product. (If the diagnosis was made prior to 2010, a diagnosis meeting the 1987 ACR classification criteria is acceptable)
* Active RA characterised by DAS28-CRP (disease activity score based on 28 joints and c-reactive protein) equal to or above 4.5 and at least five tender and five swollen joints (can be the same joints) of the 28 joint count
* Concomitant treatment with MTX above or equal to 15 mg/week for at least 4 months prior to screening, with stable dose of between or equal to 15 mg/week and 25 mg/week for at least 6 weeks prior to screening (MTX doses between 7.5 and 12.5 mg/week are allowed, if patient had intolerance to 15 mg/week)
* Biologic naïve subjects or subjects having been treated with biologics for RA (biologic experienced) provided they meet one of the following criteria: a. Reason for discontinuation of biologic therapy was intolerance (e.g., unable to receive recommended doses or achieve adequate treatment duration because of drug related side effects), b. Discontinued biologic therapy for other reasons than lack of efficacy (primary or secondary failure) or intolerance (e.g., drug holiday)

Exclusion Criteria:

* Body mass index (BMI) below or equal to 18.0 or above or equal to 38.0 kg/m^2
* Subjects with rheumatic autoimmune disease other than RA, or significant systemic involvement secondary to RA (including but not limited to vasculitis, pulmonary fibrosis, or Felty's syndrome). Subjects with secondary Sjögren's syndrome or stable hypothyroidism are eligible
* Any active or ongoing bacterial infections within 4 weeks prior to randomisation, unless treated and resolved with appropriate therapy (e.g., simple urinary tract infection)
* Any history of recurrent infections or conditions predisposing to chronic infections (e.g., bronchiectasis, chronic osteomyelitis)
* History of severe systemic fungal infection within the past 12 months prior to screening unless treated and resolved with appropriate therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2012-09; Primary Completion 2013-08 (Actual); Study Completion 2013-08 (Actual)

PRIMARY OUTCOMES:
Change in disease activity score based on 28 joints and c-reactive protein (DAS28-CRP) | Week 0, week 12

SECONDARY OUTCOMES:
ACR20/50/70 (20%, 50% or 70% improvement of ACR (American College of Rheumatology) score from baseline) | Week 12
Incidence of adverse events (AEs) | Up to week 24
Incidence of antibodies against NNC0114-0006 | Up to Week 24
Terminal serum half-life (t½) | After second dose administration at week 6
Change in serum levels of total interleukin-21 (IL-21) | Up to week 12
Change in Health Assessment Questionnaire - Disability Index score (HAQ-DI) | Week 0, week 12

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (27):
- Bulgaria (3):
  - Novo Nordisk Investigational Site, Plovdiv
  - Novo Nordisk Investigational Site, Sevlievo
  - Novo Nordisk Investigational Site, Sofia
- Hungary (4):
  - Novo Nordisk Investigational Site, Budapest
  - Novo Nordisk Investigational Site, Debrecen
  - Novo Nordisk Investigational Site, Szikszó
  - Novo Nordisk Investigational Site, Veszprém
- Novo Nordisk Investigational Site, Riga, Latvia
- Poland (7):
  - Novo Nordisk Investigational Site, Bialystok
  - Novo Nordisk Investigational Site, Bydgoszcz
  - Novo Nordisk Investigational Site, Bytom
  - Novo Nordisk Investigational Site, Elblag
  - Novo Nordisk Investigational Site, Katowice
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Warsaw
- Russia (6):
  - Novo Nordisk Investigational Site, Kazan'
  - Novo Nordisk Investigational Site, Kursk
  - Novo Nordisk Investigational Site, Moscow
  - Novo Nordisk Investigational Site, Skt Petersburg
  - Novo Nordisk Investigational Site, Skt. Petersburg
  - Novo Nordisk Investigational Site, Yaroslavl
- Serbia (2):
  - Novo Nordisk Investigational Site, Belgrade
  - Novo Nordisk Investigational Site, Niška Banja
- Spain (4):
  - Novo Nordisk Investigational Site, A Coruña
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Elche
  - Novo Nordisk Investigational Site, Seville

REFERENCES:
- [Result] Canete J, Leszczynski P, Riisbro R, Frederiksen K. Efficacy and safety of NNC0114-0006, an anti-IL-21 monoclonal antibody, in patients with active rheumatoid arthritis. Arthritis and Rheumatology; 66 (10 (Supplement)): Abstract 947
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com